CLINICAL TRIAL: NCT00286078
Title: Precision Implantable Stimulator for Migraine (PRISM) Study- Occipital Nerve Stimulation (ONS) for Migraine
Brief Title: Treatment for Migraines With an Implantable Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EI0105
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Migraine
Keywords: Headache; Migraine; Refractory; Chronic; Pain
MeSH Terms: conditions — Migraine Disorders; Headache; Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Active occipital nerve stimulation (stimulation on)
  Interventions: Device: Precision
- Control (Sham Comparator): Sham occipital nerve stimulation from activation to 12 weeks post-activation. Active occipital nerve stimulation from 12 weeks post-activation on.
  Interventions: Device: Precision

INTERVENTIONS:
Device: Precision — Implantable neurostimulator

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an implantable device for difficult to treat migraine. There are a significant number of patients who have drug refractory migraine and alternative therapies are needed.

ELIGIBILITY:
Key Inclusion Criteria:

* Be diagnosed with multiple migraines per month of moderate to severe intensity;
* Be refractory to medication;
* Be an appropriate candidate for the surgical procedures required for this study;
* Be willing and able to comply with all study related procedures;
* Be capable of reading and understanding patient information materials and giving written informed consent.

Key Exclusion Criteria:

* Have onset of migraine after age 50;
* Have a significant psychiatric disorder;
* Have previously been treated with occipital nerve stimulation;
* Have had an injection of botulinum toxin in the head or neck within 6 months prior to enrollment;
* Have previously undergone destructive ganglionectomy affecting C2/C3 occipital and/or trigeminal distribution or have an occipital blockade or radio frequency procedure currently in effect;
* Have a condition currently requiring or likely to require the use of MRI or diathermy;
* Have an active implantable device;
* Have participated in any drug or device trial in the last 4 weeks or plan to participate in any other study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lipton, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (15):
- United States (15):
  - Mile High Research Center, Denver, Colorado
  - The New England Center for Headache, Stamford, Connecticut
  - Walton Rehabilitation Hospital, Augusta, Georgia
  - Rush Pain Center, Chicago, Illinois
  - Diamond Headache Clinic, Chicago, Illinois
  - New England Regional Headache Center, Worcester, Massachusetts
  - Headache Care Center, Springfield, Missouri
  - Headache Specialists, Las Vegas, Nevada
  - Albert Einstein College of Medicine - Montefiore Headache Unit, The Bronx, New York
  - The Neurological Clinic, Portland, Oregon
  - Thomas Jefferson University - Jefferson Headache, Philadelphia, Pennsylvania
  - Nashville Neuroscience Group, Nashville, Tennessee
  - Research Center, Fort Worth, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Swedish Pain & Headache Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 179 subjects signed consent, 39 subjects screen failed, and 140 eligible subjects were randomized (1 subject was later excluded).
Period: Overall Study
Arm/Group | Treatment | Control
Started | 72 | 68
12 Weeks | 63 | 62
Completed | 40 | 34
Not Completed | 32 | 34

BASELINE CHARACTERISTICS:
Population: 1 subject excluded from analysis because HIPAA authorization was not obtained; randomized to active group, received percutaneous trial only
Groups:
- Treatment: Stimulation on
  Precision: Implantable neurostimulator
- Control: Sham Stimulation up to 12 weeks post-activation. Actual Stimulation from 12 weeks post-activation on.
  Precision: Implantable neurostimulator
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 71 | 68 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (11.2) | 43.8 (11.9) | 42.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 57 | 117
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United States | 71 | 68 | 139

OUTCOME MEASURES:

1. Primary Outcome: Migraine Frequency at 12 Weeks
Description: Change from baseline in migraine days/month at 12 weeks
Time Frame: Baseline and 12 weeks
Population: Modified Intent to Treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 63 | 62
days | -5.5 (8.7) | -3.9 (8.2)

2. Primary Outcome: Frequency of Adverse Event
Description: Cumulative frequency of adverse events from randomization to 26 weeks
Time Frame: 26 weeks
Measure: Number; unit: events
Arm/Group | Treatment | Control
Number analyzed (Participants) | 71 | 68
events | 276 | 284

ADVERSE EVENTS:
Time Frame: Safety data was collected through the 12 year follow up visit.
Arm/Group | Treatment | Control
Serious Adverse Events (participants affected / at risk) | 33/72 | 19/68
Other Adverse Events (participants affected / at risk) | 68/72 | 63/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=72) | Control (N=68)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (2) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 6 (7) | 2 (3)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Congestive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse Drug Reaction (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Implant Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Septic Embolus (Infections and infestations) | 1 (1) | 0 (0)
Stitch Abscess (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Device Lead Damage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug Toxicity (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protusion (Musculoskeletal and connective tissue disorders) | 1 (5) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Intracranial Venous Sinus Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Migraine without Aura (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Completed Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Conversion Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Subclavian Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arnold-Chiari Malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=72) | Control (N=68)
Nausea (Gastrointestinal disorders) | 16 (18) | 9 (12)
Vomiting (Gastrointestinal disorders) | 6 (7) | 2 (3)
Implant site pain (General disorders) | 10 (14) | 16 (17)
Therapeutic product ineffective (General disorders) | 46 (67) | 44 (66)
Bronchitis (Infections and infestations) | 3 (3) | 6 (6)
Nasopharyngitis (Infections and infestations) | 7 (8) | 5 (5)
Sinusitis (Infections and infestations) | 7 (9) | 10 (17)
Inappropriate device stimulation of tissue (Injury, poisoning and procedural complications) | 24 (30) | 9 (10)
Incision site complication (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Incision site pain (Injury, poisoning and procedural complications) | 5 (5) | 8 (9)
Medical device pain (Injury, poisoning and procedural complications) | 4 (4) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (10)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (9)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 10 (10)
Headache (Nervous system disorders) | 14 (22) | 9 (14)
Migraine (Nervous system disorders) | 6 (12) | 11 (13)
Insomnia (Psychiatric disorders) | 7 (7) | 4 (4)
Oedema Peripheral (General disorders) | 4 (4) | 2 (2)
Device Migration (Injury, poisoning and procedural complications) | 4 (4) | 4 (6)
Medical device complication (Injury, poisoning and procedural complications) | 5 (8) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Paresthesia (Nervous system disorders) | 6 (6) | 3 (3)
Tremor (Nervous system disorders) | 1 (1) | 4 (5)
Depression (Psychiatric disorders) | 1 (1) | 4 (5)
Insomnia (Psychiatric disorders) | 7 (8) | 6 (7)
Hypertension (Vascular disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No